CLINICAL TRIAL: NCT06277882
Title: Efficacy and Durability of Hepatitis A Vaccination in Patients With Advanced Fibrosis and Cirrhosis: A Randomized-controlled Trial
Brief Title: Efficacy and Durability of Hepatitis A Vaccination in Patients With Advanced Fibrosis and Cirrhosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Associate professor, Faculty of Medicine, Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Si 067/2024
Record Dates: First submitted 2024-02-10; First posted 2024-02-26 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Cirrhosis; Hep A; Vaccination
Keywords: Cirrhosis; HAV; Hepatitis A; HAV vaccine
MeSH Terms: conditions — Fibrosis; Hepatitis A | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive 3 dose (Experimental): Receiving the intensive 3-dose regimen of the Havrix hepatitis A vaccine, administered at months 0, 1, and 6.
  Interventions: Biological: HAVRIX
- Standard 2 dose (Active Comparator): Receiving the standard 2-dose regimen of the Havrix hepatitis A vaccine, administered at months 0, and 6.
  Interventions: Biological: HAVRIX

INTERVENTIONS:
Biological: HAVRIX — intramuscular injections
  Other Names: HAV vaccine

SUMMARY:
The hepatitis A virus (HAV) is a significant global public health concern. The hepatitis A virus is transmitted primarily by the faecal-oral route, leading to acute hepatitis. Symptoms include low-grade fever, anorexia, jaundice, and typically resolve without complications.

However, HAV infection in patients with chronic liver disease, especially those over 50 years old, may result in more severe outcomes, including fulminant hepatitis, with a higher mortality rate compared to the general population

HAV vaccination is a cornerstone of prevention, especially in high-risk groups. Currently, there is a recommendation to vaccinate patients with chronic liver disease against HAV infection. However, these patients often have compromised immune responses, leading to lower vaccine efficacy compared to the general population.

The goal of this randomized controlled trial is to compare the efficacy and safety of the standard 2-dose (0, 6 months) hepatitis A vaccination regimen with an intensive 3-dose (0, 1, 6 months) schedule in patients with advanced fibrosis and cirrhosis.

The main questions it aims to answer are:

* Compared the seroconversion rate of the standard 2-dose (0, 6 months) hepatitis A vaccination regimen versus the intensive 3-dose (0, 1, 6 months) hepatitis A vaccination regimen in patients with advanced fibrosis and cirrhosis.
* Compared the antibody levels against the hepatitis A virus (Anti-HAV IgG) of the standard 2-dose (0, 6 months) hepatitis A vaccination regimen versus the intensive 3-dose (0, 1, 6 months) hepatitis A vaccination regimen in patients with advanced fibrosis and cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed advance fibrosis (F3) or cirrhotic (F4) status (radiologic finding or liver stiffness measurement or pathological report)
* Negative anti-HAV IgM, IgG at baseline

Exclusion Criteria:

* Positive anti-HAV IgG at baseline
* Autoimmune hepatitis
* Current hepatocellular carcinoma
* Active other malignancies
* Presence of antibodies against Human Immunodeficiency Virus
* Received immunosuppressive drugs
* Pregnancy or lactation
* Decompensated cirrhosis with MELD ≥ 15
* Chronic illness or bedridden patient who cannot travel to hospital
* Lack of consent to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Post-vaccination serological response rate | At 7 months after complete vaccine administration
  To compare the seroconversion response rate at month 7
  Subjects are considered as being seroconversion if they were initially seronegative and become seropositive

SECONDARY OUTCOMES:
Post-vaccination serological response | At 30 days after first dose administration
  To compare the seroconversion response rate at month 1
  Subjects are considered as being seroconversion if they were initially seronegative and become seropositive
Post-vaccination serological response | At 1 year after first dose administration
  To compare the seroconversion response rate at 1 year
  Subjects are considered as being seroconversion if they were initially seronegative and become seropositive
Anti-hepatitis A Virus (HAV) antibody at month 1 | At 30 days after first dose administration
  To compare Anti-HAV IgG level obtained with two different vaccination schemes against HAV in advance fibrosis and cirrhotic patients
Anti-hepatitis A Virus (HAV) antibody at month 7 | At 7 months after complete vaccine administration
  To compare Anti-HAV IgG level obtained with two different vaccination schemes against HAV in advance fibrosis and cirrhotic patients
Anti-hepatitis A Virus (HAV) antibody at 1 year | At 1 year after first dose administration
  To compare Anti-HAV IgG level obtained with two different vaccination schemes against HAV in advance fibrosis and cirrhotic patients

CONTACTS AND LOCATIONS:
Overall Officials: Watcharasak Chotiyaputta, Asso Prof, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

REFERENCES:
- [Result] Advisory Committee on Immunization Practices (ACIP); Fiore AE, Wasley A, Bell BP. Prevention of hepatitis A through active or passive immunization: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2006 May 19;55(RR-7):1-23. PMID 16708058
- [Result] Keeffe EB. Is hepatitis A more severe in patients with chronic hepatitis B and other chronic liver diseases? Am J Gastroenterol. 1995 Feb;90(2):201-5. PMID 7847285
- [Result] Webb GW, Kelly S, Dalton HR. Hepatitis A and Hepatitis E: Clinical and Epidemiological Features, Diagnosis, Treatment, and Prevention. Clin Microbiol Newsl. 2020 Nov 1;42(21):171-179. doi: 10.1016/j.clinmicnews.2020.10.001. Epub 2020 Oct 22. PMID 33110280
- [Result] Lemon SM, Ott JJ, Van Damme P, Shouval D. Type A viral hepatitis: A summary and update on the molecular virology, epidemiology, pathogenesis and prevention. J Hepatol. 2017 Sep 5:S0168-8278(17)32278-X. doi: 10.1016/j.jhep.2017.08.034. Online ahead of print. PMID 28887164
- [Result] Noor MT, Manoria P. Immune Dysfunction in Cirrhosis. J Clin Transl Hepatol. 2017 Mar 28;5(1):50-58. doi: 10.14218/JCTH.2016.00056. Epub 2017 Mar 10. PMID 28507927
- [Result] Arguedas MR, McGuire BM, Fallon MB. Implementation of vaccination in patients with cirrhosis. Dig Dis Sci. 2002 Feb;47(2):384-7. doi: 10.1023/a:1013734525348. PMID 11855555
- [Result] Wigg AJ, Wundke R, McCormick R, Muller KR, Ramachandran J, Narayana SK, Woodman RJ. Efficacy of High-Dose, Rapid, Hepatitis A and B Vaccination Schedules in Patients With Cirrhosis. Clin Gastroenterol Hepatol. 2019 May;17(6):1210-1212.e1. doi: 10.1016/j.cgh.2018.08.047. Epub 2018 Aug 23. PMID 30144521
- [Result] Ioannou GN. HCC surveillance after SVR in patients with F3/F4 fibrosis. J Hepatol. 2021 Feb;74(2):458-465. doi: 10.1016/j.jhep.2020.10.016. Epub 2020 Dec 7. PMID 33303216